CLINICAL TRIAL: NCT01888757
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover, Oral Bioequivalence Study in Healthy, Adult, Human Subjects Under Fed Conditions.
Brief Title: Lamotrigine Extended-Release Tablets 50 mg Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 718/09
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: Bioequivalence; Lamotrigine Extended Release; crossover
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine Extended Release Tablets (Experimental): Lamotrigine Extended Release Tablets, 25 mg, 50 mg, 100 mg, 200 mg and 300 mgof Dr. Reddy's Laboratories Limited
  Interventions: Drug: Lamotrigine
- LAMICTAL XR (Active Comparator): (containing Lamotrigine)Extended Release tablets 50 mg of GlaxoSmithKline Research Triangle Park, NC
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine Extended Release Tablets, 25mg, 50mg, 100mg, 200mg and 300 mg
  Other Names: LAMICTAL XR

SUMMARY:
This is an open label, randomised, balanced, two-treatment, two-period, two-sequence, single dose, crossover, oral bioequivalence study.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover, oral bioequivalence study of Lamotrigine Extended Release tablets 50 mg of Dr. Reddy's Laboratories Limited, India comparing with that of LAMICTAL XR(containing Lamotrigine) Extended Release tablets 50mg of GlaxoSmithKline Research Triangle Park, NC in healthy, adult, human subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects were selected based on the following inclusion criteria:

* Provide written informed consent.
* Must be healthy, adult, human beings within 18 and 45 years of age (both inclusive) weighing at least 50 kg.
* Having a body mass index between 18.5 and 24.9 (both inclusive), calculated as weight in Kg/height in m 2.
* Must be of normal health as determined by medical history, physical examination and laboratory investigation performed within 28 days prior to the commencement of the study. (Laboratory values must be within normal limits or considered by the physician / investigator to be of no clinical significance).
* Female Subjects

  * Of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
  * Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria The subjects were excluded based on the following criteria during screening and during the study:

* Incapable of understanding the informed consent.
* Systolic blood pressure less than 90 mm of Hg or more than 140 mm of Hg.
* Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg.
* Oral temperature is below 95.0°F or above 98.6°F.
* Pulse rate below 50/min or above 100/min.
* History of hypersensitivity or idiosyncratic reaction to investigational drug product or any other related drugs or its ingredients.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.
* Consumption of grapefruit for the past ten days prior to the check-in, in each period.
* Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking during sample collection period.
* Habit of tobacco chewing.
* Habit of alcoholism and difficulty in abstaining from alcohol during the sample collection period.
* Difficulty in abstaining from xanthine containing food or beverages (like tea, coffee, chocolates and cola drinks) during the sample collection period.
* Intake of over the counter (OTC) or prescribed medications and enzyme modifying medication or systemic medication for the last 30 days before dosing.
* Clinically significant abnormalities and / or with significant diseases.
* Confirmed positive in alcohol screening.
* Confirmed positive in urine cotinine test.
* Confirmed positive in selected drug of abuse.
* Participated in any other clinical investigation using experimental drug/donated blood in past 90 days before the date of start of study.
* Confirmed positive in urine pregnancy test. xx. Female detected to be pregnant, breast feeding or who is likely to become pregnant during the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Area under curve(AUC) | Predose (0.00) and 1.00, 2.00, 3.00, 4.50, 6.00, 7.50, 9.00, 10.50, 12.00, 13.50, 15.00, 16.50, 18.00, 20.00, 22.00, 24.00, 26.00, 30.00, 36.00, 48.00, 72.00, 96.00, 120.00, 144.00 and 168.00 post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Vimal Teja P, Dr., Principal Investigator — Bioserve Clinical Research Private Limited,
Locations (1):
- Bioserve Clinical Research Private Limited, Bālānagar, Hyderabad, India